CLINICAL TRIAL: NCT00002028
Title: A Treatment IND (Investigational New Drug) Protocol for the Use of Videx (2',3'-Dideoxyinosine, ddI) in Patients With Acquired Immunodeficiency Syndrome (AIDS) or AIDS- Related Complex (ARC) Who Are Intolerant to Zidovudine (Retrovir)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 040A; 454-999-001
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2007-08-16 (Estimated); Status verified 2007-08

CONDITIONS: HIV Infections
Keywords: Didanosine; Drugs, Investigational; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Zidovudine
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Didanosine

INTERVENTIONS:
Drug: Didanosine

SUMMARY:
The objective of this treatment IND protocol is to make didanosine (ddI) available to patients with HIV infection (suffering from AIDS related complex (ARC) or AIDS) who have developed documented intolerance to zidovudine (AZT) and cannot enter a Phase II ddI program due to protocol exclusion or geographic location.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* Concomitant medications for the treatment of AIDS or ARC (including aerosolized pentamidine).
* Phenytoin, but with caution.
* Note:
* Extreme caution should be exercised in the use of ddI in any patient receiving concomitant therapies, particularly those receiving other nucleosides (e.g. ganciclovir), drugs with toxicities similar to those observed with ddI (list included under concomitant medications section of protocol), and other drugs with significant toxicities, including many drugs used for treatment of major opportunistic infections.

Patients must:

- Have a diagnosis of AIDS or be symptomatic, HIV positive, and have a CD4 cell count < 200 cells/mm3.

Be intolerant to zidovudine (AZT) therapy. Not be suitable for study entry into the phase II didanosine (ddI) study by reason of inclusion or exclusion criteria or by reason of geographic location.

Be able to provide signed informed consent (parent/guardian as appropriate). Be available for monthly follow-up while taking ddI. Meet baseline lab criteria within 14 days prior to initial drug dosing.

Note:

* Extreme caution should be exercised in the use of ddI in any patient receiving concomitant therapies, particularly those receiving other nucleosides (e.g., ganciclovir), drugs with toxicities similar to those observed with ddI (list included under concomitant medications section of protocol), and other drugs with significant toxicities, including many drugs used for treatment of major opportunistic infections.

Caution should also be exercised in a patient having intractable diarrhea or patients following a low-sodium diet. Physicians caring for patients must perform clinical and laboratory evaluations every 7 - 10 days for the first 2 months of ddI therapy. All high-risk patients (for example, patients with preexisting disorders of body systems known to be adversely affected by ddI, particularly those with a history of peripheral neuropathy, pancreatitis, seizure disorder, cardiac abnormalities, gout, and significant elevations of liver function test results), must have clinical and laboratory evaluations performed every 10 days and results submitted to Bristol-Myers Squibb on the case report forms provided.

Prior Medication:

Allowed:

* Anti-emetic medication.
* Required:
* Zidovudine (AZT).

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* Malignancy likely to require chemotherapy in the first 3 months of ddI treatment.
* Acute pancreatitis.
* A poorly controlled seizure disorder.
* Grade B or greater peripheral neuropathy.

Concurrent Medication:

Excluded:

* Zidovudine (AZT).
* Chemotherapy in the first 3 months of ddI treatment.

Patients with the following are excluded:

* Malignancy likely to require systemic chemotherapy in the first 3 months of ddI treatment.
* Acute pancreatitis.
* A poorly controlled seizure disorder.
* Grade B or greater peripheral neuropathy.

Prior Medication:

Excluded within 15 days of study entry:

* Any antiretroviral drug except zidovudine (AZT).

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- Bristol - Myers Squibb Co, Princeton, New Jersey, United States

REFERENCES:
- [Background] Connolly KJ, Allan JD, Fitch H, Jackson-Pope L, McLaren C, Canetta R, Groopman JE. Phase I study of 2'-3'-dideoxyinosine administered orally twice daily to patients with AIDS or AIDS-related complex and hematologic intolerance to zidovudine. Am J Med. 1991 Nov;91(5):471-8. doi: 10.1016/0002-9343(91)90182-w. PMID 1659189